CLINICAL TRIAL: NCT00679965
Title: A Randomized, Double-Blind, Vehicle-Controlled, Multi-Center Study to Evaluate the Safety and Efficacy of Topically Applied AN2690 2.5%, 5.0%, and 7.5% Solutions vs. Vehicle for the Treatment of Adult Subjects With Onychomycosis of the Great Toenail
Brief Title: Study of Different Doses of a Novel Treatment for Onychomycosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AN2690-ONYC-200; C3371001 (Other: Alias Study Number)
Record Dates: First submitted 2008-05-15; First posted 2008-05-19 (Estimated); Last update posted 2018-12-12 (Actual); Status verified 2018-12

CONDITIONS: Distal, Subungual Onychomycosis
Keywords: Onychomycosis; Fungal Nail
MeSH Terms: conditions — Onychomycosis | interventions — tavaborole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group 1 (Experimental): AN2690 Solution, 2.5%
  Interventions: Drug: AN2690, 2.5%
- Group 2 (Experimental): AN2690 Solution: 5%
  Interventions: Drug: AN2690, 5%
- Group 3 (Experimental): AN2690 Solution, 7.5%
  Interventions: Drug: AN2690, 7.5%
- Group 4 (Placebo Comparator): AN2690 Solution Vehicle
  Interventions: Drug: AN2690 Solution Vehicle

INTERVENTIONS:
Drug: AN2690, 2.5% — Once daily application for 90 days and 3 x weekly for 90 days
  Arms: Group 1
Drug: AN2690, 5% — Once daily application for 90 days and 3 x weekly for 90 days
  Arms: Group 2
Drug: AN2690, 7.5% — Once daily application for 90 days and 3 x weekly for 90 days
  Arms: Group 3
Drug: AN2690 Solution Vehicle — Once daily application for 90 days and 3x weekly for 90 days
  Arms: Group 4

SUMMARY:
The purpose of the study is to determine the safety and efficacy of 2.5%, 5.0%, and 7.5% AN2690 Solutions compared to the vehicle alone in the treatment of distal, subungual onychomycosis of the great target toenail.

DETAILED DESCRIPTION:
The intent is for all subjects to complete a 180 day treatment period consisting of 90 consecutive days of once daily treatment with their assigned study treatment followed by an additional 90 days of three times weekly dosing, even if the treated toenail(s) is evaluated as a "complete responder" prior to the end of treatment 180 day treatment period.

At the end of the 180-Day treatment period, subjects who remain in the study will be classified as complete responders, partial responders, or non-responders. All complete or partial responders will continue to be followed for an additional 180 days until the last evaluation for inclusion in the final analysis.

Periodic efficacy and local tolerance evaluations of the test medication will be performed of the target great toenail and all other treated toenails. KOH wet mounts and fungal cultures from the treatment-targeted great toenail will be performed on the same schedule.

Subjects will also be queried for adverse events and evaluated for application site reactions. Clinical laboratory assessment for safety will be made at Screening, periodically throughout the study, and upon premature discontinuation from the study.

ELIGIBILITY:
Inclusion Criteria:

1. Witnessed, signed informed consent approved by Institutional Review Board/Ethics Committee.
2. Male or female subjects of any race at least 18 years of age but not older than 65 years of age.
3. Subjects with a diagnosis of onychomycosis of at least one great toenail and with a positive KOH wet mount and a positive fungal culture for a dermatophyte.
4. Onychomycosis involving 20-60% of the affected great toenail as determined at baseline (Day 1) by visual inspection after the nail has been trimmed.
5. The combined thickness of the distal nail plate and the associated hyperkeratotic nail bed < 3 mm.
6. Affected great toenail to be treated is capable of re-growth as documented by history or recent observation of at least 2 mm of growth.
7. Normal or not clinically significant screening safety labs.

Exclusion Criteria:

1. Females of childbearing potential not using a highly effective method of birth control (e.g. implants, injectables, combined oral contraceptives, some intrauterine contraceptive devices) during the study.
2. Diabetes mellitus requiring treatment other than diet and exercise.
3. Subjects with chronic moccasin type of T. pedis.
4. Subjects with a history of having failed any previous topical antifungal therapy for their onychomycosis.
5. Subjects unwilling to refrain from the use of nail cosmetics such as clear and/or colored nail lacquers from the screening visit until the end of the study.
6. Subjects that have not undergone the specified washout period(s) for the following topical preparations or subjects who require the concurrent use of any of the following topical medications:

   1. Topical antifungal applied to the feet (does not include antifungals for treatment of T. pedis during the study): 4 weeks
   2. Anti-inflammatories, corticosteroids, topical immunomodulators: 2 weeks
7. Subjects that have not undergone the specified washout period(s) for the following systemic medications or subjects who require the concurrent use of any of the following systemic medications:

   1. Corticosteroids (including intramuscular injections): 2 weeks
   2. Antifungals for treatment of onychomycosis or any systemic antifungal with known activity against dermatophyte: 24 weeks
   3. Systemic immunomodulators: 4 weeks
8. Treatment of any type for cancer within the last 6 months.
9. History of any significant internal disease.
10. Subjects with a medical history of current or past psoriasis of the skin and/or nails.
11. Concurrent lichen planus.
12. Subjects who are known to be allergic to any of the test product(s) or any components in the test product(s) or history of hypersensitivity or allergic reactions to any of the study preparations as described in the Investigator's Brochure.
13. Nail or anatomic abnormalities of the toe, e.g., genetic nail disorders, primentary disorders, onychogryphosis, trauma to the nail(s) to be treated.
14. AIDS or AIDS related complex.
15. History of street drug or alcohol abuse.
16. Any subject not able to meet the study attendance requirements.
17. Subjects who have participated in any other trial of an investigational drug or device within 60 days prior to enrollment or participation in a research study concurrent with this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2006-02-28 (Actual); Primary Completion 2007-07-31 (Actual); Study Completion 2007-07-31 (Actual)

PRIMARY OUTCOMES:
Clinical evidence of complete great toenail clearance or at least fungal-clear great toenail growth ("complete" = 5mm; "partial" = 2mm), plus a negative fungal culture from the treatment-targeted great toenail. | Day 180

SECONDARY OUTCOMES:
Absence of signs and symptoms of onychomycosis plus a negative fungal culture & negative KOH from the treatment-targeted toenail. | Day 360

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (9):
- Mexico (9):
  - Unidad de Investigación en Salud (UIS), Chihuahua City
  - Hospital "Dr. Angel Leaño", Guadalajara
  - Instituto Dermatologico Jalisciense, Guadalajara
  - Centro Dermatologico Pascua, Mexico City
  - CIF-BIOTEC Medica Sur., Mexico City
  - IMIC, Mexico City
  - Hospital Universitario Dr. José Eleuterio González, Monterrey
  - MIRC / OCA Hospital, Monterrey
  - ISSEMYM, Toluca